CLINICAL TRIAL: NCT04836390
Title: A Phase II Pilot Study of Donor-Derived Ex-Vivo Expanded Natural Killer Cell Infusions in Children and Young Adults With High Risk Acute Myeloid Leukemia Receiving Myeloablative HLA-Haploidentical Hematopoietic Cell Transplant: A Multicenter Pediatric Transplantation and Cellular Therapy Consortium (PTCTC) Study
Brief Title: Donor-Derived Ex-Vivo Expanded Natural Killer Cell Infusions in Children and Young Adults With High Risk Acute Myeloid Leukemia Receiving Myeloablative HLA-Haploidentical Hematopoietic Cell Transplant
Acronym: EXCEL
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Pulsipher (Other)
Collaborators: Nationwide Children's Hospital (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Michael Pulsipher, Sponsor-Investigator, Pediatric Transplantation & Cellular Therapy Consortium
Organization: Pediatric Transplantation & Cellular Therapy Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-20-00314
Record Dates: First submitted 2021-03-18; First posted 2021-04-08 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): All subjects will receive NK infusions.
  Interventions: Drug: Donor-Derived Ex-Vivo Expanded Natural Killer Cell Infusions

INTERVENTIONS:
Drug: Donor-Derived Ex-Vivo Expanded Natural Killer Cell Infusions — Peripheral blood (PB) ≤ 450 mL and based on donor weight (minimum 10 ml/kg) will be drawn from the HLA-haploidentical donor at least 16 days before the scheduled day of transplant (Day 0). HaploNK cells will be manufactured from the PB of the donor after co-culture with irradiated feeder cells (IFC) as described in Section 2.4. The recipients will receive three NK cell infusions on Day-1, Day+7 (± 1 day) and Day+42 (up to Day+90) from day of transplant (Day 0).

SUMMARY:
This is a Phase II pilot study to determine the efficacy of three fixed dose (1 x 108/kg) infusions of ex-vivo expanded human leukocyte antigen (HLA)-haploidentical donor natural killer (NK) cells (haploNK) in children and young adults with high risk acute myeloid leukemia (AML) undergoing HLA-haploidentical hematopoietic cell transplant (haploHCT) with a busulfan and cyclophosphamide-based myeloablative conditioning regimen and post-transplant cyclophosphamide (PTCy) for graft versus host disease (GVHD) prophylaxis. The investigators will also demonstrate the feasibility of performing this trial in a multi-center study.

The investigators hypothesize that the infusion of haploNK in this setting will facilitate immune reconstitution and decrease relapse rates and infectious complications without increasing GVHD, resulting in improved survival as compared to recent historical cohorts of haploHCT without NK cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 25 years at time of enrollment
* High-risk AML, as defined by one of the following:
* AML in CR1 (defined as <5% blasts in BM by morphology and flow cytometry) having at least one of these high-risk features:
* Mutations associated with high risk disease (Appendix A). Other high-risk features not explicitly stated in Appendix A can be considered after discussion/approval with the protocol chair/team
* MRD-positive at the end of Induction I chemotherapy (defined as flow cytometry ≥ 0.1% blasts)
* AML in ≥CR2 (defined by <5% blasts in BM by morphology and flow cytometry)
* Recovery from prior cycle of chemotherapy as defined by an absolute neutrophil count ≥ 500/mm3
* AML secondary to select germline marrow failure disorders (with exception of Fanconi Anemia) may be eligible but require approval from Protocol Chairs prior to enrollment.
* Performance status ≥70% (Lansky for <16 years; Karnofsky for ≥16 years)
* Adequate major organ system function as demonstrated by:
* Renal: Creatinine clearance (CrCl) ≥60 mL/min/1.73m2 by Cockcroft-Gault formula, Schwartz formula, or nuclear GFR study (Table 3)
* Hepatic: Total bilirubin <2 mg/dL (unless due to Gilbert syndrome) and ALT and AST < 5x ULN
* Cardiac: LVEF at rest ≥50% or SF ≥27% (by MUGA or ECHO)
* Pulmonary: DLCO, FEV1, and FVC ≥ 50% of predicted corrected for hemoglobin. For patients <7 years of age or those unable to perform PFTs: O2 Sat >92% on room air by pulse oximetry and on no supplemental O2 at rest
* The patient, patient's parent, guardian, or legal representative can provide written informed consent

Exclusion Criteria:

* Active extramedullary disease
* Unresolved/ongoing and serious viral, bacterial, or fungal infection despite appropriate treatment
* Positive pregnancy test in a female of child-bearing potential (FCBP)
* Inability to comply with medical therapy or follow-up
* Prior allogeneic transplant
* Patients with Fanconi Anemia and Down syndrome

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
1-year RFS | 1 year
  The proportion and corresponding 95% exact binomial CI of patients who are relapse-free at 1-year from day of transplant (Day 0)

SECONDARY OUTCOMES:
Number of functional donor-derived NK cells generated from the device | 2 years
  Product manufacturing failure is defined as inability to generate sufficient NK cell product due to failure to meet release criteria or insufficient cells for at least one full dose (≤10^8/NK cells/kg ABW).
GVHD incidence | 2 years
  The incidence of Grade II- IV aGVHD (Day +100) and cGVHD (Day+180, +1 year), opportunistic infections (+1 year), and OS (+1 year and +2 year).
KIR ligand-ligand mismatch | 2 years
  The presence of KIR ligand-ligand mismatch between HLA-haploidentical donor and host and the impact on relapse rate.
Incidence of mixed donor chimerism | 2 years
  Mixed donor chimerism is defined as >5%, but <95%, donor cells detected. Full donor chimerism is defined as >95% donor.
Cumulative incidence of neutrophil engraftment | 2 years
  The cumulative incidence of neutrophil engraftment from the time of transplant will be estimated using the cumulative incidence function with death and relapse prior to engraftment as the competing risk. The definition of neutrophil engraftment is a post-nadir ANC > 500/mm3 for three consecutive laboratory values obtained on different days. The first of the three days will be designated as the day of neutrophil recovery.
Cumulative incidence of platelet engraftment | 2 years
  The cumulative incidence of platelet engraftment from the time of transplant will be estimated using the cumulative incidence function with death and relapse prior to engraftment as the competing risk. The definition of platelet engraftment is sustained platelet count > 20,000/mm3 with no platelet transfusions in the preceding seven days. The first of three consecutive measurements on different days will be designated as the day of initial platelet recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Pulsipher, MD, Study Director — Children's Hospital Los Angeles
Locations (13):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Washington University, St. Louis, St Louis, Missouri
  - New York Medical College, Valhalla, New York
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data analysis and protocol can be made available to researchers upon request after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for an additional 2-3 years.
Access Criteria: Contact Principal Investigator